CLINICAL TRIAL: NCT07090655
Title: A Phase 1, Randomized, Double-blind, Placebo-controlled, Single-ascending-dose Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of Subcutaneous and Intravenous Injections of Budoprutug (TNT119) in Normal Healthy Volunteers
Brief Title: A Phase 1 Study of Budoprutug (TNT119) Subcutaneous and Intravenous Injections in Normal Healthy Volunteers
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Climb Bio, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Basic Science
Other Study IDs: TNT119-NHV-101
Record Dates: First submitted 2025-07-21; First posted 2025-07-29 (Actual); Last update posted 2025-08-20 (Actual); Status verified 2025-08

CONDITIONS: Healthy Volunteers
Keywords: healthy; volunteer

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Budoprutug (Experimental): Subcutaneous (SC) injection or IV administration of budoprutug
  Interventions: Drug: Budoprutug
- Placebo (Placebo Comparator): Placebo solution to be administered at a matching volume
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Budoprutug — Subcutaneous or IV administration
  Other Names: TNT119
  Arms: Budoprutug
Drug: Placebo — Placebo comparator
  Arms: Placebo

SUMMARY:
The main objective is to assess the safety and tolerability of subcutaneous and intravenous injection forms of budoprutug in healthy volunteers.

DETAILED DESCRIPTION:
Budoprutug is a humanized, immunoglobulin (Ig) G1 monoclonal antibody that selectively binds to CD19 and is projected to deplete targeted cells through antibody-dependent cellular cytotoxicity. This Phase 1, randomized, double-blind, placebo-controlled, single-ascending-dose study is designed to evaluate the safety, tolerability, pharmacokinetics (PK), and pharmacodynamics (PD) of budoprutug administered subcutaneously (SC) in adult normal healthy volunteers (NHVs). To assess the bioavailability of the SC formulation, one cohort will receive a single intravenous (IV) dose of budoprutug. Approximately 38 participants will be enrolled across four dose cohorts, including three SC dose levels and one IV comparator group.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adult males and females aged 18-60 years
* Body mass index (BMI) between 18 and 32 kg/m² and weight between 45 and 110 kg
* Clinically normal medical history, physical exam, ECG, and laboratory results (or abnormalities deemed not clinically significant)
* Willing and able to comply with study procedures and provide informed consent
* Women of childbearing potential must use highly effective contraception and have negative pregnancy tests
* Men must use contraception and refrain from sperm donation for 6 months post-dose
* Completion of a 2-dose primary COVID-19 vaccination series and at least 1 booster dose, as well as influenza vaccination (within 12 months)

Exclusion Criteria:

* Prior treatment with investigational drugs within 30 days or 5 half-lives
* History of hypogammaglobulinemia or significant allergic reactions
* Recent infections, including serious local/systemic infections or opportunistic infections
* Positive tests for HIV, hepatitis B/C, syphilis, or tuberculosis
* Use of tobacco (>2 cigarettes/day), alcohol abuse, or recreational drugs
* Recent live vaccination (within 21 days) or any non-live vaccine (within 14 days)

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 38 (Estimated)
Dates: Start 2025-08-11 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Safety and Tolerability of Single Ascending Doses of budoprutug in Healthy Participants | Day 57
  Incidence of treatment-emergent adverse events
Incidence of infusion-related reactions (IRRs) for IV administration | Day 57
  Number of infusion-related reactions
Incidence of injection site reactions (ISRs) for SC administration | Day 57
  Number of injection site reactions

SECONDARY OUTCOMES:
Maximum Observed Plasma Concentration (Cmax) | Day 57
  Measurement of the maximum observed plasma concentration.
Time to Maximum Observed Concentration (Tmax) | Day 57
  Measurement of the time to maximum observed concentration.
Area Under the Curve (AUC) | Day 57
  Measurement of the area under the drug concentration-time curve.
Terminal Half-Life (T1/2) | Day 57
  Measurement of the terminal half-life in days.
Bioavailability (F) | Day 57
  Relative absorption of SC vs IV budoprutug (%).

CONTACTS AND LOCATIONS:
Locations (1):
- Nucleus Network Brisbane, Brisbane, Australia